CLINICAL TRIAL: NCT00314392
Title: Effect of Participant Gender, Experimenter Gender, and Drug-Related Information on Placebo Analgesia
Brief Title: Gender, Pain, and Placebo Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: The Research Council of Norway (Other); University of Tromso (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Placebo
Record Dates: First submitted 2006-04-11; First posted 2006-04-13 (Estimated); Last update posted 2008-02-06 (Estimated); Status verified 2008-02

CONDITIONS: Experimental Pain
Keywords: Experimental pain; Placebo analgesia; Heart rate variability; Skin conductance

INTERVENTIONS:
Behavioral: Information (behavior)

SUMMARY:
The response to standard pain stimuli in males and females is investigated, together with the effect of informing participants about the effect of a painkiller. Physiological response to pain is recorded.

DETAILED DESCRIPTION:
The social context in which pain is reported has been found to modulate pain. Specifically, male participants reporting pain to female observers report significantly lower pain levels compared to male participants reporting to male observers. Female participants seem less affected by social context. This is a methodological problem in the study of pain and has consequences in the development of new drugs, and for pain research in general.

The present study has two aims: To investigate whether social context affects also the placebo response to pain, i.e. the reduced pain often observed after administration of a an inert substance the participants believes to be a painkiller. It is hypothesized that placebo analgesia will be larger in males reporting pain to females. Secondly, heart rate variability and skin conductance, measures of parasympathetic and sympathetic activity, will be recorded, to investigate if social context affects not only pain report, but also pain response.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years, healthy

Exclusion Criteria:

* pregnant, earlier serious disease or injury,

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2006-09; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Pain report, heart rate variability, skin conductance

SECONDARY OUTCOMES:
Subjective arousal

CONTACTS AND LOCATIONS:
Overall Officials: Magne Arve Flaten, PhD, Principal Investigator — University of Tromso
Locations (1):
- University Hospital of North Norway, Tromsø, Troms, Norway